CLINICAL TRIAL: NCT01023594
Title: Comparison of Feasibility Between Internal and External Pancreatic Drainage in Pancreaticoduodenectomy: Prospective Randomized Study
Brief Title: Comparison of Feasibility Between Internal and External Pancreatic Drainage in Pancreaticoduodenectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Sun-Whe Kim, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-0908-040-290
Record Dates: First submitted 2009-11-30; First posted 2009-12-02 (Estimated); Last update posted 2015-09-15 (Estimated); Status verified 2015-09

CONDITIONS: Pancreatic Fistula
Keywords: Pancreatic fistula; Pancreatic leakage; Pancreatoduodenectomy; Pancreatic stent
MeSH Terms: conditions — Pancreatic Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- External stent (Active Comparator): Feeding tube insert at pancreatojejunostomy site as a stent. And stent tube is brought out through jejunal loop below the hepaticojejunostomy site and abdominal wall.
  Interventions: Procedure: Pancreatic stent
- Internal stent (Active Comparator): short(5cm)internal stent insertion at pancreatojejunostomy site
  Interventions: Procedure: Pancreatic stent

INTERVENTIONS:
Procedure: Pancreatic stent — Feeding tube insert at pancreatojejunostomy site as a stent. And then 1) tube is brought out through jejunal loop below the hepaticojejunostomy site and abdominal wall(external stent)or 2) tube is cut short (5cm length) and left in situ with fixating suture. In external stent group, tube will be removed about 1 months after operation.

SUMMARY:
Pancreatic fistula is one of the most serious complication after pancreatoduodenectomy. To reduce pancreatic fistula, many authors recommend pancreatic stent in pancreatojejunostomy. There are two distinct methods of pancreatic stent insertion: internal stent and external stent. There was few studies comparing these methods in preventing pancreatic fistula. Furthermore, its long-term effect was not known enough. The purpose of this study is to determine which is the best method in preventing pancreatic fistula and to investigate its long term clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* patient who have malignant or benign disease which needs pancreatoduodenectomy
* patient age: ≥20 and ≤85

Exclusion Criteria:

* patient who had chemotherapy or radiotherapy previous to operation.
* patient who had severe comorbid disease(cardiac, pulmonary, cerebrovascular)
* patient who had past medical history of chronic pancreatitis.
* pancreatic stent size <1mm or >5mm

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328 (Estimated)
Dates: Start 2010-01; Primary Completion 2014-01 (Actual); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
evidence of pancreatic fistula confirmed by serum and drain amylase | within the first 7 days after surgery

SECONDARY OUTCOMES:
pancreatic endocrine and exocrine function by blood test, stool exam (steatorrhea) and computed tomography (CT) volumetry | within the first 1 year after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Sun-Whe Kim, M.D., Study Chair — Seoul National University Hospital
Locations (8):
- South Korea (8):
  - Center for Liver Cancer, National Cancer Center, Goyang-si, Gyeonggi-do
  - Department of Surgery, Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Department of Surgery, Seoul National University Hospital, Seoul, Seoul
  - Department of Surgery, Samsung Medical Center, Seoul
  - Department of Surgery, Korea University Guro Hospital, Seoul
  - Department of Surgery, Seoul National University Boramae Hospital, Seoul
  - Department of Surgery, Chung-ang University College of Medicine, Seoul
  - Department of Surgery, Gangnam Severance Hospital, Seoul

REFERENCES:
- [Background] Bassi C, Dervenis C, Butturini G, Fingerhut A, Yeo C, Izbicki J, Neoptolemos J, Sarr M, Traverso W, Buchler M; International Study Group on Pancreatic Fistula Definition. Postoperative pancreatic fistula: an international study group (ISGPF) definition. Surgery. 2005 Jul;138(1):8-13. doi: 10.1016/j.surg.2005.05.001. PMID 16003309
- [Background] Lowy AM, Lee JE, Pisters PW, Davidson BS, Fenoglio CJ, Stanford P, Jinnah R, Evans DB. Prospective, randomized trial of octreotide to prevent pancreatic fistula after pancreaticoduodenectomy for malignant disease. Ann Surg. 1997 Nov;226(5):632-41. doi: 10.1097/00000658-199711000-00008. PMID 9389397
- [Background] Butturini G, Daskalaki D, Molinari E, Scopelliti F, Casarotto A, Bassi C. Pancreatic fistula: definition and current problems. J Hepatobiliary Pancreat Surg. 2008;15(3):247-51. doi: 10.1007/s00534-007-1301-y. Epub 2008 Jun 6. PMID 18535760
- [Background] Poon RT, Fan ST, Lo CM, Ng KK, Yuen WK, Yeung C, Wong J. External drainage of pancreatic duct with a stent to reduce leakage rate of pancreaticojejunostomy after pancreaticoduodenectomy: a prospective randomized trial. Ann Surg. 2007 Sep;246(3):425-33; discussion 433-5. doi: 10.1097/SLA.0b013e3181492c28. PMID 17717446
- [Background] Roder JD, Stein HJ, Bottcher KA, Busch R, Heidecke CD, Siewert JR. Stented versus nonstented pancreaticojejunostomy after pancreatoduodenectomy: a prospective study. Ann Surg. 1999 Jan;229(1):41-8. doi: 10.1097/00000658-199901000-00005. PMID 9923798
- [Background] Kamoda Y, Fujino Y, Matsumoto I, Shinzeki M, Sakai T, Kuroda Y. Usefulness of performing a pancreaticojejunostomy with an internal stent after a pancreatoduodenectomy. Surg Today. 2008;38(6):524-8. doi: 10.1007/s00595-007-3662-x. Epub 2008 May 31. PMID 18516532
- [Background] Ohwada S, Tanahashi Y, Ogawa T, Kawate S, Hamada K, Tago KI, Yamada T, Morishita Y. In situ vs ex situ pancreatic duct stents of duct-to-mucosa pancreaticojejunostomy after pancreaticoduodenectomy with billroth I-type reconstruction. Arch Surg. 2002 Nov;137(11):1289-93. doi: 10.1001/archsurg.137.11.1289. PMID 12413321
- [Background] Imaizumi T, Hatori T, Tobita K, Fukuda A, Takasaki K, Makuuchi H. Pancreaticojejunostomy using duct-to-mucosa anastomosis without a stenting tube. J Hepatobiliary Pancreat Surg. 2006;13(3):194-201. doi: 10.1007/s00534-005-1037-5. PMID 16708294
- [Background] Kim SW, Youk EG, Park YH. Comparison of pancreatogastrostomy and pancreatojejunostomy after pancreatoduodenectomy performed by one surgeon. World J Surg. 1997 Jul-Aug;21(6):640-3. doi: 10.1007/s002689900286. PMID 9230663
- [Background] Winter JM, Cameron JL, Campbell KA, Chang DC, Riall TS, Schulick RD, Choti MA, Coleman J, Hodgin MB, Sauter PK, Sonnenday CJ, Wolfgang CL, Marohn MR, Yeo CJ. Does pancreatic duct stenting decrease the rate of pancreatic fistula following pancreaticoduodenectomy? Results of a prospective randomized trial. J Gastrointest Surg. 2006 Nov;10(9):1280-90; discussion 1290. doi: 10.1016/j.gassur.2006.07.020. PMID 17114014
- [Derived] Jang JY, Chang YR, Kim SW, Choi SH, Park SJ, Lee SE, Lim CS, Kang MJ, Lee H, Heo JS. Randomized multicentre trial comparing external and internal pancreatic stenting during pancreaticoduodenectomy. Br J Surg. 2016 May;103(6):668-675. doi: 10.1002/bjs.10160. Epub 2016 Apr 4. PMID 27040594